CLINICAL TRIAL: NCT05219721
Title: An Exploratory Study of Fully Human Anti-GPRC5D Chimeric Antigen Receptor T Cells (CAR-GPRC5D) in Patients With Relapsed/Refractory Multiple Myeloma or Plasma Cell Leukemia
Brief Title: A Study of CAR-GPRC5D in Patients With Relapsed/Refractory Multiple Myeloma or Plasma Cell Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chunrui Li (Other)
Collaborators: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chunrui Li, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD138CI001
Record Dates: First submitted 2022-01-04; First posted 2022-02-02 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Relapsed/Refractory Multiple Myeloma; Plasma Cell Leukemia
Keywords: CAR-T; GPRC5D
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell

STUDY DESIGN:
Intervention Model Description: This study pre-defined three dose levels of 1.0×10^6 CAR-T/Kg, 2.0×10^6 CAR-T/Kg, 3.0×10^6 CAR-T/Kg. Each dose level will enroll 3-6 subjects, and the estimated total number of subjects will be 9-18. This study is to observe the characteristics of dose-limiting toxicity (DLT), pharmacokinetics, pharmacodynamics, and immunogenicity of CAR-GPRC5D in different dose groups. And to preliminarily observe the efficacy in small samples of patients with R/R MM or Plasma cell leukemia and confirm the recommended phase II dose (RP2D).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-GPRC5D cells (Experimental): After lymphodepletion, CAR-GPRC5D will be administered as a single infusion.
  Interventions: Drug: CAR-T (CAR-GPRC5D)

INTERVENTIONS:
Drug: CAR-T (CAR-GPRC5D) — CAR-GPRC5D (RD118) is an individualized, gene-modified autologous T-cell immunotherapy product targeting GPRC5D that identifies and eliminates malignant and normal cells expressing GPRC5D. The CAR structure comprises a fully human single-domain antibody fragment (VHH) targeting GPRC5D, fused with intracellular co-stimulatory (4-1BB) and activation (CD3ζ) signaling domains.

SUMMARY:
This study is a single-center, open-label, dose-exploration study to observe the safety and efficacy of different doses of CAR-GPRC5D in patients with R/R MM or plasma cell leukemia.

DETAILED DESCRIPTION:
Apheresis will be performed to manufacture CAR-GPRC5D chimeric antigen receptor (CAR) modified T cells. Bridging therapy is allowed between apheresis and lymphodepletion. Lymphodepletion with fludarabine and cyclophosphamide was performed for three consecutive days. Then, subjects will receive a single dose infusion of CAR-GPRC5D at 1.0, 2.0, or 3.0 x 10^6 CAR+ T cells/Kg. Subjects will be followed in the study for a minimum of 2 years after infusion. Long-term follow-up for lentiviral vector safety will be followed for up to 15 years after infusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy all the following criteria to be enrolled in the study:

  1. age 18 to 75 years old, male or female.
  2. Subjects have had at least 3 prior lines of therapy including chemotherapy based on proteasome inhibitors (PIs) and immunomodulatory agents (IMiDs).

     According to the International Myeloma Working Group (IMWG) consensus (2016) standard on multiple myeloma, the disease has recurred, progressed or is refractory, or according to the IMWG consensus (2013) standard on plasma cell leukemia (Appendix 4), the disease appears relapse, progress or refractory;
  3. Evidence of cell membrane GPRC5D expression, as determined by a validated immunohistochemistry (IHC) or flow cytometry of tumor tissue (e.g., bone marrow biopsies, or plasmacytoma).
  4. The subjects should have measurable disease based on at least one of the following parameters:

     The proportion of primitive immature or monoclonal plasma cells detected by bone marrow cytology, bone marrow biopsy, or flow cytometry is ≥ 10%.

     Serum M-protein ≥ 0.5 g/dL. Urine M-protein ≥ 200 mg/24 hrs. For those whose Serum or Urine M-protein does not meet the measurable criteria but the light chain type, serum free light chain (sFLC) : involved sFLC level ≥ 10mg/dL (100 mg/L) provided serum FLC ratio is abnormal.

     In subjects with extramedullary myeloma, if there are no other evaluable lesions, require extramedullary lesions with a maximum diameter of ≥2cm
  5. ECOG performance score 0-2.
  6. Estimated life expectancy ≥ 12 weeks.
  7. Subjects should have adequate organ function:

     * Hematology: Absolute neutrophil count (ANC) ≥1×10^9 /L (prior use of growth factor support is permitted, but subjects must not have received supportive treatment within 7 days prior to laboratory examination); absolute lymphocyte count (ALC) ≥0.3×10^9 /L; platelets ≥40×10^9 /L (subjects must not have received blood transfusion support within 7 days prior to laboratory examination); hemoglobin ≥60 g/L (subjects must not have received transfusion of red blood cells [RBC] within 7 days prior to laboratory examination; the use of recombinant human erythropoietin is permitted).
     * Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×upper limit of normal (ULN); total serum bilirubin ≤ 1.5×ULN.
     * Renal function: Creatinine clearance rate (CrCl) calculated according to Cockcroft-Gault formula ≥ 40 ml/min.
     * Coagulation function: Fibrinogen ≥ 1.0 g/L; activated partial thromboplastin time (APTT) ≤ 1.5×ULN, prothrombin time (PT) ≤1.5×ULN.
     * SpO2 > 91%.
     * Left ventricular ejection fraction (LVEF) ≥ 50%.
  8. The subject and his/her spouse agree to use an effective contraceptive tool or medication (excluding safety period contraception) for one year from the date of the subject's informed consent to the date of CAR T cell infusion.
  9. Subject must sign the informed consent form approved by ethics board in person before starting any screening procedure.

     Exclusion Criteria:
* The presence of any of the following will exclude a subject from enrollment:

  1. Subjects who are known to have GVHD or need long-term immunosuppressive therapy.
  2. Subjects have received any anti-cancer treatment as follows:

     monoclonal antibody for treating multiple myeloma within 21 days before leukapheresis, or cytotoxic therapy or proteasome inhibitors within 14 days before leukapheresis, or immunomodulatory agents within 7 days before leukapheresis. or anti-tumor treatments other than those listed above within 30 days before leukapheresis.
  3. Subjects who were receiving a used therapeutic dose of corticosteroid treatment (defined as prednisone or equivalent > 20mg) within 7 days prior to screening, except for physiological alternatives, inhalation, or topical use.
  4. Subjects with hypertension that cannot be controlled by medication.
  5. Subjects with serious heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (NYHA classification ≥III), and severe arrhythmias.
  6. Subjects with systemic diseases that the investigator determined to be unstable include, but are not limited to, severe liver and kidney or metabolic diseases requiring medical treatment.
  7. Subjects with second malignancies in addition to MM within the past 5 years before the screening, exceptions to this criterion: successfully treated cervical carcinoma in situ and non-metastatic basal or squamous cell skin carcinoma, local prostate cancer after radical surgery, and ductal carcinoma in situ of the breast after radical surgery.
  8. Subjects with a history of organ transplantation.
  9. Subjects have received major surgery within 2 weeks prior to leukapheresis or plan to receive surgery during the study or within 2 weeks after the study treatment (excluding local anesthesia).
  10. Subjects participated in another interventional clinical study 1 months before signing the informed consent (ICF);
  11. Subjects with any uncontrolled active infection needed to receive systemic therapy within 7 days before leukapheresis collection (excluding # CTCAE grade 2 urogenital infection and upper respiratory infection).
  12. Positive for any of the following tests:

      * Hepatitis B virus (HBV) surface antigen (HBsAg) or hepatitis B core antibody-positive and detectable HBV DNA in peripheral blood
      * Hepatitis C virus (HCV) antibody and hepatitis C virus RNA in peripheral blood
      * Human immunodeficiency virus (HIV) antibody
      * Cytomegalovirus (CMV) DNA
      * Treponema Pallidum antibody
  13. Pregnant or lactating women.
  14. Subjects with mental illness or consciousness disorder or disease of the central nervous system
  15. Other conditions that researchers consider inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) by dose group | 28 days after CAR-T cell infusion
  Dose limiting toxicity will be assessed after infusion in each dose group
Type and incidence of adverse events (AEs) and serious adverse events (SAEs) by dose group | 2 years after CAR-T cell infusion
  Calculate type and incidence of adverse events (AE), serious adverse event (SAE), including those happened after lymphodepletion and after infusion, those related to study drug and lymphodepletion, or those that led to withdrawal from the study. They will also be aggregated by systematic organ classification (SOC), preferred term (PT), and severity

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years after CAR-T cell infusion
  The percentage of participants who achieved PR or better response.
Overall survival (OS) | 2 years after CAR-T cell infusion
  OS is measured from the date of the initial infusion of CAR-GPRC5D to the date of the participant's death
Duration of response (DOR) after administration | 2 years after CAR-T cell infusion
  DOR will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria
Progression-free survival (PFS) | 2 years after CAR-T cell infusion
  The time from the start of CAR-GPRC5D treatment for the participants to the first time of disease progression or death for any reason
Time to response (TTR) | 2 years after CAR-T cell infusion
  The time interval between the first treatment of CAR-GPRC5D and the time of first recording of sCR or CR or VGPR or PR of the participants
Time to complete Response (TTCR) | 2 years after CAR-T cell infusion
  Time from CAR-GPRC5D infusion to first documentation of complete response of the participants
Percentage of Participants With Negative Minimal Residual Disease (MRD) | 2 years after CAR-T cell infusion
  MRD negative rate is defined as the proportion of participants who achieve MRD negative status by the respective time point
Pharmacokinetics - Cmax | 2 years after CAR-T cell infusion
  The maximum transgene level at Tmax
Pharmacokinetics - Tmax | 2 years after CAR-T cell infusion
  Time to peak transgene level
Pharmacokinetics - AUC0-28days | 2 years after CAR-T cell infusion
  Area under the curve of CAR-T cells from time zero to Day 28
Pharmacokinetics - AUC0-90days | 2 years after CAR-T cell infusion
  Area under the curve of CAR T cells from time zero to Day 90
PD endpoints - the level of free CAR-GPRC5D | 2 years after CAR-T cell infusion
  The content of free CAR-GPRC5D in peripheral blood will be detected at each time point
PD endpoints - the levels of CAR-T-related serum cytokines | 2 years after CAR-T cell infusion
  The concentration levels of CAR-T-related serum cytokines (such as IL-6) will be detected at each time point
Health-related quality of life assessment | 2 years after CAR-T cell infusion
  HRQoL will be assessed by the European Organization for Cancer Research and Treatment Quality of Life Questionnaire (EORTC-QLQ-C30)
Evaluation of lymphocyte subsets | 2 years after CAR-T cell infusion
  Lymphocyte subsets will be assessed by FACS
Levels of immunoglobulins | 2 years after CAR-T cell infusion
  Immunoglobulins in peripheral blood will be assessed to monitor changes

OTHER OUTCOMES:
Positive rate of human anti-CAR antibody | 2 years after CAR-T cell infusion
  The levels of human anti-CAR antibody of participants will be detected
Number of Participants with replication competent lentivirus (RCL) | 2 years after CAR-T cell infusion
  Number of participants exhibiting anti-drug antibodies for CAR-GPRC5D will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Chunrui Li, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Pan M, Wang D, Xu J, Jin S, Wang Y, Tao Y, Liu Y, Ouyang W, Weng X, Yi H, Huang Y, Cao X, Li S, Zhang F, Zhang W, Li C, Mi JQ. Fully Human anti-GPRC5D CAR T-Cell Therapy RD118 Induces Durable Remissions in Relapsed/Refractory Multiple Myeloma. Blood. 2025 Oct 21:blood.2025030559. doi: 10.1182/blood.2025030559. Online ahead of print. PMID 41118600